CLINICAL TRIAL: NCT04393883
Title: A Randomized, National Multicenter Clinical Study Comparing Pembrolizumab With Maintenance Therapy Every 3 Weeks and Every 6 Weeks for First-line Treatment of PD-L1 ≥1% Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study With Pembrolizumab for Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Guangzhou Medical University (Other); Southern Medical University, China (Other); Beijing Sino-Japan Friendship Hospital (Unknown); First Hospital of China Medical University (Other); Changhai Hospital of the Second Military Medical University (Unknown); Jiangsu People's Hospital (Unknown); Qilu Hospital of Shandong University (Other); Tongji Hospital (Other); Xijing Hospital Affiliated to the Fourth Military Medical University (Unknown); Xiangya Hospital of Central South University (Other); West China Hospital (Other); The Second Affiliated Hospital of the Army Medical University (the Third Military Medical University) - Xinqiao Hospital (Unknown); Zunyi Medical College (Other); The Second Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR2019001206
Record Dates: First submitted 2020-05-06; First posted 2020-05-19 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-04

CONDITIONS: Non-small-lung-cell Cancer, NSCLC; Pembrolizumab
Keywords: (Non-small-lung-cell cancer, NSCLC) subjects,Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard maintenance programme group (Experimental): pembrolizumab 200mg, every 3 weeks, for a total of 2 years of follow-up and follow-up for 1 year;
  Interventions: Drug: A) Standard maintenance programme group, pembrolizumab 200mg, every 3 weeks, for a total of 2 years of follow-up and follow-up for 1 year;
- Improvement maintenance programme group, (Experimental): pembrolizumab 200mg, every 6 weeks, for a total of 2 years of follow-up and 1 year follow-up;
  Interventions: Drug: B) Improvement maintenance programme group, pembrolizumab 200mg, every 6 weeks, for a total of 2 years of follow-up and 1 year follow-up;

INTERVENTIONS:
Drug: A) Standard maintenance programme group, pembrolizumab 200mg, every 3 weeks, for a total of 2 years of follow-up and follow-up for 1 year; — (A) Standard maintenance programme group, pembrolizumab 200mg, every 3 weeks, for a total of 2 years of follow-up and follow-up for 1 year;
  Arms: Standard maintenance programme group
Drug: B) Improvement maintenance programme group, pembrolizumab 200mg, every 6 weeks, for a total of 2 years of follow-up and 1 year follow-up; — (B) Improvement maintenance programme group, pembrolizumab 200mg, every 6 weeks, for a total of 2 years of follow-up and 1 year follow-up;
  Arms: Improvement maintenance programme group,

SUMMARY:
This study is a randomized, national multicenter clinical study ，which is designed to compare the efficacy of the safety and efficacy of treatment every 3 weeks or 6 weeks in (Non-small-cell-cell cancer, NSCLC) subjects without systematic treatment， who used Pembrolizumab after 6 cycles of combined chemotherapy， estimated with stable efficacy (CR, PR, and SSD) .

In this study, subjects will be randomly assigned to the following two groups according to a 1:1 ratio:

(A) Standard maintenance programme group, pembrolizumab 200mg, every 3 weeks, for a total of 2 years of follow-up and follow-up for 1 year; (B) Improvement maintenance programme group, pembrolizumab 200mg, every 6 weeks, for a total of 2 years of follow-up and 1 year follow-up;

DETAILED DESCRIPTION:
This study is a randomized, national, multicenter clinical study aimed at non-small-cell lung cancer (NSCLC) subjects with PD-L1 ≥ 1% who have not previously received systematic treatment After comparing Pembrolizumab alone or Pembrolizumab combined with chemotherapy for 6 cycles, after the efficacy evaluation was stable (CR, PR, and SD), the safety and clinical efficacy of maintenance therapy every 3 weeks and every 6 weeks were compared. The eligible subjects in this study will be randomly assigned into the following two groups according to the 1: 1 ratio:

(A) Standard maintenance program group, namely Pembrolizumab 200mg, every 3 weeks, a total of 2 years of treatment, followed up for 1 year; (B) Modified maintenance program group, namely Pembrolizumab 200mg, every 6 weeks, a total of 2 years of treatment, followed up for 1 year;

During the course of the trial treatment, if the subject develops disease (the first PD), the researcher will decide whether to continue the medication according to the patient's situation and communicate with the patient, and decide whether to unblind according to the specific situation, as follows: After the first PD of the subject, the researcher decides whether to continue the treatment with the original regimen according to the disease state of the subject. At least 4 weeks later, the tumor is evaluated again. If the tumor progresses again (the second PD), the subject's study treatment ends and the follow-up period is entered; if there is no progress, the original regimen is continued. If the subjects decide to continue to use Pembrolizumab-related treatment after PD, they must meet the corresponding indicators of the enrollment and exclusion criteria of this study:

1. No clinical symptoms and signs of significant disease progression (including worsening of laboratory examination results).
2. ECOG's physical performance score is stable.
3. Critical anatomical sites (such as spinal cord compression) did not see rapid disease progression or tumor progression requiring urgent alternative medical interventions.
4. The main organ function meets the corresponding laboratory indexes in the inclusion and exclusion criteria of this study.
5. The subject must sign the "Informed Consent for Continued Medication after the First Disease Progression".

The primary end point of this study was to compare the incidence of treatment-related grade 3-5 adverse events between the standard maintenance group and the modified maintenance group. The secondary end point was descriptive analysis of progression-free survival and overall survival. Using RECIST 1.1 as the evaluation standard, the independent imaging evaluation committee (IRRC) conducted the evaluation. For the first time to evaluate PD, regardless of whether they continue to study treatment after progression, the date of the first PD evaluated by IRRC will be used for all statistical analysis containing progress information.

ELIGIBILITY:
Inclusion Criteria:

-

1. Volunteer for clinical research, fully understand, inform and sign informed consent forms (Informed Consent Form, ICF), willing to follow and be able to complete all trial procedures. 2. 18 to 75 years old (with critical values) when signing ICF. 3. Hemology diagnostics of phase IV (AJCC Version 8) NSCLC that cannot be surgicalor-able or radiotherapy. 4. No known EGFR sensitivity mutations or ALK, ROS1 gene rearrangement; 5. Patients have never received systemic treatment throughout the body for phase IV NSCLC. 6. The end of non-systematic anti-tumor therapy is not only 2 weeks from the end of the study drug, and the treatment-related AE is restored to CTCAE 4.03 to level 1 (except for level 2 hair loss). 7. Within 4 weeks prior to randomization, at least one measurable target lesions assessed by irRC in accordance with RECIST 1.1 requirements. 8. Patients must provide the required tumor tissue for PD-L1 expression level determination, and PD-L1 is 1%. Note: Samples of tumor tissue fixed by Formalin within 6 months prior to the first study of the drug use are recommended. Paraffin encapsulated tumor specimens (preferred) or unstained newly cut continuous tissue slices (preferred anti-stripping slides). A relevant pathological report of the above specimen sits must also be provided. Freshly collected specimens, excision, hollow needle core biopsy, excision, cut, stamping or clamp biopsy are all within acceptable range (preferred newly acquired tissue). Needle-absorbing samples (i.e., samples that lack a complete tissue structure only provide cell suspension and/or cell smears), brush samples, cell precipitation samples from chest or celiac fluidares are not accepted. The organization sample requirements are detailed in the laboratory operating manual. 9. The ECOG PS score for 7 days prior to the first drug use of the study drug was 0 or 1. 10. After 6 cycles of combination chemotherapy with Pembrolizumab 200mg Q3W or Pembrolizumab 200mg Q3W immunotherapy, the efficacy was assessed as CR, PR, SD. 11. The expected lifetime is 12 weeks. 12. The main organ function sits well, i.e. meets the following criteria (no blood transfusion, albumin, recombinant human platelet production or csphylitosin (CSF) treatment within 14 days prior to the first drug use in this study): 13. Organ function is normal:

1. White blood cells s.0 x 109/L
2. Absolute Neutlyte Granucyte Count (ANC) s2.0 x 109/L
3. Platelet count: 100 x 109/L
4. Hemoglobin s 90 g/L
5. Creatine s 1.5 x ULN;
6. Total bilirubin s 1.5 x ULN (except Gilbert syndrome, total bilirubin 3.0 mg/dL);
7. AST (SGOT) is 2.5 x ULN, for patients with liver metastiars, s.5 x ULN;
8. ALT (SGPT) is 2.5 x ULN, for patients with liver metastasis, s.5 x ULN;
9. Alkaline phosphatase is 3 times the normal upper limit;
10. Clotting function: activated part of the clotting enzyme time (APTT) s1.5 x ULN, clotting enzyme raw time (PT) or international standardized ratio (INR) s1.5 x ULN;
11. Female patients must meet one of the following:

(1) menopause (defined as having no menstruation for at least 1 year and no other reason for confirmation other than menopause); (2) sterilization performed (removal of the ovaries and/or uterus); (3) Fertility, but must meet: Serum pregnancy tests must be negative within 7 days of randomization and agree to use 1% annual failure rate of contraception or to maintain abstinence (avoiding heterosexual intercourse) (at least 120 days after the signing of an informed consent form to the last time the drug was administered) (1% annual failure rate of contraceptive methods including bilateral tubal ligation, male sterilization, correct use of ovulation-suppressing hormones, release of intrauterine and intrauterine devices) and intrauterine devices. 12) Male patients must meet the requirement to consent to abstinence (avoiding heterosexual intercourse) or to take contraception, provided that when the partner is a woman of childbearing age or who is pregnant, male patients must maintain abstinence or use condom contraception to prevent exposure to the embryo during treatment and for at least 150 days after the end of administration of the drug. Regular abstinence (e.g. calendar days, ovulation periods, basic body temperature or late-stage contraception) and in vitro ejaculation are substandard methods of contraception.

Exclusion Criteria:

1. Histological type is small cell lung cancer or mixed tumors with small cell lung cancer, neuroendocrine cancer components. 2. Within 5 years or at the same time, there are other active malignancies. Cured limited tumors, such as skin base cell carcinoma, skin squamous carcinoma, superficial bladder cancer, prostate in situ cancer, cervical in situ cancer, breast in situ cancer, etc. can be included in the group. 3. A patient who is prepared to undergo or have received an organ or bone marrow transplant in the past. 4. Chest fluid, cardiac fluid or ascites that cannot be controlled by appropriate intervention. 5. Known or screened examinations found in patients with active central nervous system (CNS) metastasis and/or cancerous meningitis. However, the following patients are allowed to join the group: 1) Asymptomatic brain metastasis patients (i.e. no brain metastasis caused by the development of sexual central nervous system symptoms, do not require glucocorticoid therapy, and the size of the lesions of 1.5cm) can participate, but the disease site needs to be regularly examined for brain imaging. 2) In patients with after treatment of brain metastasis, and brain metastasis lesions are stable for at least 1 month, there is no new or enlarged evidence of brain metastasis, and glucocorticoids are discontinued for 3 days before administration. Stable brain metastasis should be determined prior to the first drug use. 6. Surgery and/or radiotherapy fail to cure spinal cord compression. 7. Obviously hemorrhagic, combined patients with venous syndrome. 8. Myocardial infarction and poor control of arrhythmia (including QTc interstitallated men with a period of 450 ms and female s470 ms) occurred in the first six months prior to the first drug use (QTc interstitallator is calculated using the Fridericia formula). 9. In accordance with NYHA Standard III- IV level cardiac insufficiency or cardiac color super-examination: LVEF (left ventricular blood score) 50%. 10. Poor control of hypertension (i.e. systolic pressure (BP) of 150 mmHg and/or diastolic pressure of 100 mmHg), has previously appeared high blood pressure risk or hypertension encephalopathy. 11. The patient had CTCAE 4.03 peripheral neuropathy level 2. 12. Human immunodeficiency virus (HIV) infection. 13. He suffers from active tuberculosis. 14. Past and current patients with interstitial pneumonia, dust lung, radiocopmedy, drug-related pneumonia, severe lung function, etc., may interfere with the monitoring and treatment of suspected drug-related pulmonary toxicity. 15. Patients have known active or suspected autoimmune diseases. Patients who are allowed to be in a stable state and do not require systemic immunosuppressants. 16. Hepatitis B (HBsAg or HBcAb tested positive and HBV-DNA tested positive), hepatitis C (hCV antibody tested positive and HCV-RNA positive). Subjects with a common infection with hepatitis B and C (HBsAg or HBcAb tested positive and HCV antibodies tested positive). 17. A live vaccine is treated within 28 days of the first drug use, but seasonal influenza is permitted, but the detoxified live flu vaccine is not allowed to be administered with nasal medication. 18. Patients who need to be treated with systemic glucocortical extrex (?10 mg/temponnison) or other immunosuppressive medications within 14 days of the first drug use or during the study. However, admission is permitted in the group where patients are allowed to use topical or inhaled glucocorticoids and adrenal corticosteroid replacement therapy at a dose of 10 mg/templiison. 19. Any active infectionthat that requires systemic anti-infection treatment occurs within 14 days of the first drug use. 20. Within 28 days of the first drug use, major surgery was undergone, and the study defined major surgery: at least 3 weeks of recovery time after surgery to be able to undergo surgery for this study. Tumor punctures or lymph node cut biopsies are allowed into the group. 21. Within 3 months of the first drug use, he received thetogenive radiation therapy. Note: Palliative radiotherapy for bone palliative radiotherapy or superficial lesions is permitted, the course of treatment is based on local standards and is completed 2 weeks prior to the first dose. Radiotherapy covering more than 30% of the bone marrow area is not permitted within 28 days of the first use. 22. Patients have previously received other antibodies/drugs against immuno-checking points, such as PD-1, PD-L1, CTLA4, etc. 23. Participating in other clinical studies, or planning to begin treatment for this study is less than 14 days from the end of the previous clinical study. 24. A history of severe allergies to any monoclonal antibody is known. 25. Pregnant or lactating women. 26. Patients are known to have a history of psychotropic substance abuse or drug abuse; 27. The researchers determined that the patient had other factors that might have caused the study to be forced to terminate in the middle.

-

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | three years
  Patients with oncological diseases have a period of time from the start of treatment to the observation of disease progression or death due to any cause

SECONDARY OUTCOMES:
objective response rate | three years
  Refers to the proportion of patients whose tumor shrinkage reaches a certain amount and remains for a certain period of time, including CR + PR cases
OS：overall survival | three years
  The time from randomization to death due to any cause. For subjects who have been lost to follow-up before death, the time of the last follow-up is usually calculated as the time of death.
Duration of mitigation (DOR) | three years
  Refers to the event that the first evaluation of the tumor is CR or PR to the first evaluation of PD or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Fen Lan, Principal Investigator — Fen lan， Kejin Yin, Chenzhi Zhou, Shaoxi Cai, Ting Yang, Gang Hou, Cong Bai, Mao Huang, LIang Dong,
Locations (1):
- Key Laboratory of Respiratory Disease of Zhejiang Province, Department of Respiratory and Critical Care Medicine, Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, 310009, China, Hangzhou, Zhejiang, China